CLINICAL TRIAL: NCT02486965
Title: Impact of a Specific Training Program on the Neuromodulation of Pain in Fibromyalgia Subjects
Acronym: DOUFISPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DOUFISPORT (RB 14.076)
Record Dates: First submitted 2015-02-26; First posted 2015-07-01 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Fibromyalgia
Keywords: VAS; thermode test; training program; 6MWT
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- training group (Experimental): The training program consists of three sessions of 45 minutes of physical activity per week for 2 years. During the first 6-9 months, two individual workouts, supervised by a physiotherapist and a session in Living.
  Depending on the capacity and exercise tolerance of the patient, patients realize the second phase of training until 2 years of the study: three exercise sessions from 45 to 60 minutes per week of which group session led by a professor of Adapted Physical Activity (APA) and 2 autonomous sessions.
  Thermal stimulation with test thermode Thermic stimulations (tonic heat pain stimulation and cold-pressor test) are used to test excitatory and inhibitory pain mechanisms
  Interventions: Device: thermode (TSA-II model); Other: Adapted Physical Activity; Other: Physical activity
- control group (Placebo Comparator): A training program supervised by physical therapists and teachers in Adapted Physical Activity, identical to the active program in its follow-up, but the intensity of the sessions is lower than that of the training group
  Interventions: Other: Adapted Physical Activity

INTERVENTIONS:
Device: thermode (TSA-II model) — thermal stimulation with test thermode
  Arms: training group
Other: Adapted Physical Activity
Other: Physical activity
  Arms: training group

SUMMARY:
Fibromyalgia affects 1.4 now 2.2% of the general population whose symptom is the presence of widespread pain in all four quadrants of the body. Currently, there is no causal treatment of fibromyalgia syndrome.

The aim of this study is the evaluation of a specific training program on controls of pain in fibromyalgia patients by balancing the stress axis.

The primary endpoint is the improvement in the Visual Analogue Scale VAS difference) measured during the test of the thermode (difference between the average VAS measured between the 10th and 40th second of P1 and the average VAS measured between the 10th and 40th of the second P3) between D0 (3rd consultation) and M24 (5th consultation - end of study visit), which will be compared in the two groups..Salivary cortisol is also tested.

DETAILED DESCRIPTION:
A specific training program under the guidance of a physiotherapist, a professor of Adapted Physical Activity (APA) and individualized whose objective is to strengthen the parasympathetic tone and modulate the reactivity of the sympathetic system and the report of the Hypothalamic-Pituitary-Adrenal (HPA) axis.This training program consists of three sessions of 45 minutes of physical activity per week for 2 years. The exercise intensity is initially very low and will be gradually increased according to your abilities and your tolerance to stress. A 6-Minute Walk Test (6MWT) will be carried out by the physiotherapist and by Professor APA, every 6 months to monitor the progression. For tracking the training program, a phone call is scheduled every week during the first 3 months, then a phone call every 15 days during the following months until the end of the study.Evaluation of neuromodulation of pain will be measured thanks to thermodeTest , experimental method implementing a tonic thermal pain using a "Peltier type Thermode" 3 cm2 model TSA II and immersion in a bath of cold water.

Participants will be randomly assigned to 2 groups, "Training" group or "Control" group.

The control group is a training program supervised by physical therapists and teachers in Adapted Physical Activity, identical to the active program in its follow-up, but the intensity of the sessions is lower.

Study schedule :

* 1st visit : screening visit at D-30
* 2nd visit : inclusion at D-7
* 3rd visit at D0
* 4st visit between M6 and M9
* 5th visit at M24

The patients included in the study will receive in addition to the training program, taking into bio-psycho-social multidisciplinary.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia is clearly established by the criteria of the American College of Rheumatology (ACR).
* Body Mass Index (BMI) between 18.5 and 24.9 kg / m² (normal weight at HAS).
* Spontaneous pain intensity greater than 3/10 on a VAS. Pain triggered by palpation must be equal to or greater than 4/10 of the EVA.
* Patients with a medical certificate to the sport.

Exclusion Criteria:

* Systemic disease, whether or not, generating pain musculoskeletal
* Heart disease, respiratory, endocrine, metabolic or neurological.
* Patients and patient pregnant lactating or planning to become pregnant within 2 years.
* Patients who have changed in the last 2 months any pharmacological treatment.
* Patients taking drugs that affect the heart rate variability
* Patients who have conditions that could affect the cortisol levels
* Patients with a psychiatric diagnosis of schizophrenia, delusional disorder and other personality disorders
* Patients taking substances affecting cortisol secretion

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Pain as assessed by Visual analog scale | baseline to 24 months

SECONDARY OUTCOMES:
salivary cortisol | baseline to 24 months
  three times : 3th visit at Day 0, 4th visit between month 6 and 9, 5th visit at month 24
heart rate variability | baseline to 24 months
  three times : 2th visit at Day -7, 4th visit between month 6 and 9, 5th visit at month 24
Fibromyalgia Impact Questionnaire (FIQ) | baseline to 24 months
Hospital Anxiety Depression Scale (HADS) | baseline to 24 months
Pressure Pain Threshold (PSS) | baseline to 24 months
International Physical Activity Questionnaire (IPAQ) | baseline to 24 months
Pittsburgh Sleep Quality Index (PSQI) | baseline to 24 months
Saint-Antoine Pain Questionnaire (SAPQ) | baseline to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gildas L'HEVEDER, Doctor, Principal Investigator — CHRU Brest
Locations (2):
- France (2):
  - CHRU Brest, Brest
  - CHU Rennes, Rennes

REFERENCES:
- [Derived] Le Fur Bonnabesse A, Cabon M, L'Heveder G, Kermarrec A, Quinio B, Woda A, Marchand S, Dubois A, Giroux-Metges MA, Rannou F, Misery L, Bodere C. Impact of a specific training programme on the neuromodulation of pain in female patient with fibromyalgia (DouFiSport): a 24-month, controlled, randomised, double-blind protocol. BMJ Open. 2019 Jan 25;9(1):e023742. doi: 10.1136/bmjopen-2018-023742. PMID 30782715